CLINICAL TRIAL: NCT00583245
Title: Optimizing Mobility in Older Adults With Knee Osteoarthritis
Brief Title: Improving Walking in Older Adults With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Neil A Segal, Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200704794; 1K23AG030945-01 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Gait training; Knee pain; Rehabilitation; Physical Therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Gait training
  Interventions: Other: Gait Training

INTERVENTIONS:
Other: Gait Training — Gait training with physical therapist 2/week for 3 months

SUMMARY:
Knee osteoarthritis (OA) accounts for a significant proportion of mobility limitations and is one of the most disabling problems facing the growing population of older adults. The long-term objective of this research is to reduce disablement of older adults with symptomatic knee OA. The principle of specificity of training indicates that exercises that closely approximate the goal functional activity are most effective in improving physical performance during that activity. Based on this principle, the specific aim of this pilot study is to design a patient-specific gait training intervention using analysis of compensatory joint moments and energy expenditure. Successful completion will inform rehabilitation for maintaining or improving mobility as well as explore the mechanism of effect.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee osteoarthritis (knee osteoarthritis diagnosed by x-ray and frequent knee symptoms)
* Age 60 or older

Exclusion Criteria:

* acute or terminal illness
* unstable cardiovascular condition or other medical conditions that may impair ability to participate such as pulmonary disease requiring the use of supplemental oxygen, neurological disease that affects gait, or lower limb musculoskeletal surgery in the past 6 months.
* Bilateral knee replacement

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Changes in functional limitation assessed by the A) Summary Performance Score which includes balance tests, timed 4-meter walk, and timed chair stand test B) Timed stair climb C) Late Life Function and Disability Instrument (LLFDI) Questionnaire | 12 weeks
Changes in the disability measure, a timed 400 meter walk | 12 Weeks
Changes in impairments assessed using the Knee and Osteoarthritis Outcome Score (KOOS) questionnaire | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil Segal, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States